CLINICAL TRIAL: NCT04999930
Title: Comparison of Clinical Efficacy and Patient's Satisfaction of Tiotropium Respimat Administration With and Without Aerochamber in Patient With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Tiotropium Respimat Administration With and Without Aerochamber Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Mohamed Faisal Abdul Hamid, Associate Professor Doctor, National University of Malaysia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FF-2019-462
Record Dates: First submitted 2021-06-18; First posted 2021-08-11 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): with aerochamber
  Interventions: Device: Aerochamber
- Group B (Experimental): without aerochamber
  Interventions: Device: Aerochamber

INTERVENTIONS:
Device: Aerochamber — efficacy and patients satisfaction
  Other Names: Tiotropium respimart

SUMMARY:
COPD patient on Tiotropium Respimart divided into two group, Group A given aerochamber and Group B without aerochamber enroll in the study for total 18 week .

DETAILED DESCRIPTION:
1. COPD patient who is on Tiotropium Respimart and other inhalers continued.
2. Those fullfill inclusion criteria will be randomized into two group.
3. To do Baseline CAT score and SGRQ questionnaires with Lung function test.
4. Assess inhaler technique with and without aerochamber.
5. Teach proper inhaler technique by templates and demonstrate to patients.
6. Group A given aerochamber and Group B without aerochamber enroll in the study for total 18 week .
7. First phase for 8 week after that 2 week of washout periode (without aerochamber both arm).
8. Then Group A without aerochamber and Group B with aerochamber continue with all inhalers for 8 week.
9. Followed up at 8th , 11th and 18th week to assess inhaler techniques ,Lung function test and do CAT score, and SGRQ questionnaire.
10. Analysis data

ELIGIBILITY:
Inclusion Criteria:

1. COPD patients under Respiratory clinic UKM follow up

   * Patients who are with stable COPD (no exacerbation past 2 months)
   * Age same and more than 40-year-old
2. Patient able to perform inhaler medication
3. Patient able to perform technically acceptable pulmonary function test

Exclusion Criteria:

1. Drug hypersensitivity
2. Bronchial Asthma
3. Significant disease that may influence patient's ability to participate in the study.
4. Unable to provide signed informed consent
5. Mental condition rendering the subject unable to understand the nature, scope and the possible consequences of the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
To compare the frequency of exacerbation (number of events ) and hospital admission (number of admissions) using tiotropium with and without aerochamber | 18 weeks
  Comparing frequency of exacerbation (number of events ) and hospital admission (number of admissions) in both groups

SECONDARY OUTCOMES:
Change of FEV1 (%) between the treatment group | 18 weeks
  Comparing differences of lung function (FEV1 %) in both groups after cross-over
Types of inhaler technique error between the group | 18 weeks
  Comparing inhaler errors in both groups based on the checklist
To assess quality of life (SGRQ questionaire) | 18 weeks
  Scores range from 0 to 100, with higher scores indicating more limitations.
To assess patients satisfaction and preference, attitudes, and perceptions about their inhalers using questionnaire | 18 weeks
  Scale of 0-5, (0-very easy, 5-hard)

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Malaysia, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No